CLINICAL TRIAL: NCT03929237
Title: When do School-aged Patients Return to School After ACL Surgery?
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: University of Michigan (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Scott Kaar, MD, Associate Professor, St. Louis University
Other Study IDs: 29979
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: ACL Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observe when return to school after surgery — Short written questionnaire asking when they returned to school and what accommodations, if any, the school made available for them

SUMMARY:
We intend to survey school aged patients following ACL surgery on when they return to school. We will analyze independent variables to determine if any relationship exists that may influence the amount of time missed.

DETAILED DESCRIPTION:
All patients undergoing ACL surgery who are enrolled in middle or high school will be recruited for study participation. Patients undergoing concomitant additional ligament surgery will be excluded. The only procedure will be to answer a short written questionnaire asking when they returned to school and what accommodations, if any, the school made available for them. This will occur at the patient's 2 week post-operative clinic visit. This clinic visit is a standard of care visit. Independent variables will be collected from the medical record and are all standard of care information routinely collected from this patient populations (age, sex, race, date of surgery, surgeon, sport played, grade, ACL surgery graft type, associated meniscal or chondral surgery, length of post-operative narcotic use, regional nerve block at the time of surgery, SANE score, IKDC score, brace used).

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction surgery
* currently enrolled in middle or high school (grades 6-12)
* Surgery occurs during the school year
* No concomitant additional ligament surgery (ie. PCL, MCL, LCL or MPFL)

Exclusion Criteria:

* patient is home schooled or in non-traditional school setting (ie. school for special needs)
* concomitant additional ligament surgery
* surgery occurs outside of the school year or on a scheduled break from school

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: School aged patients who undergo ACL reconstruction surgery during the school year
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
When return to school after surgery | 1-2 weeks post-operatively
  days from surgery to return to school

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No